CLINICAL TRIAL: NCT02190370
Title: Within Subject Design on the Efficacy of a Resources Activation Treatment Programme in Children and Adolescents With Tics
Brief Title: Efficacy of a Resources Activation Treatment on Tic-symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Manfred Doepfner, Leading psychologist at the Department of Childhood and Adolescence Psychiatry, University of Cologne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: THICS-Study 3
Record Dates: First submitted 2014-04-14; First posted 2014-07-15 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Tic-Disorder
Keywords: Tic-Disorder, Tourette-Disorder, Resources activation
MeSH Terms: conditions — Tics; Tourette Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Resources activation (Experimental): At first patients get informed about Tics in general. Through different exercises existing resources and skills are activated and strengthened. Feeling of self-esteem and self-respect are strengthened. Also the emotional awareness is strengthened. Relaxation methods are also introduced.
  Interventions: Behavioral: Resources activation

INTERVENTIONS:
Behavioral: Resources activation

SUMMARY:
The main purpose of this study is to evaluate the efficacy of a resources activation based treatment programme in children and adolescents aged 8 to 18 years with tic disorders.

DETAILED DESCRIPTION:
The main purpose of this study is to evaluate the efficacy of an intervention aimed at the activation of resources for children and adolescents with tic disorders. The activation of resources treatment programme was developed at Department of Child and Adolescent Psychiatry and Psychotherapy at the University of Cologne and is currently evaluated in different studies.

ELIGIBILITY:
Inclusion Criteria:

* 8-18 years
* Diagnosis of chronic motor or vocal Tic (F95.1) or Tourette-Syndrome (F95.2)
* YGTSS total score F95.2>13, F95.1>9
* Tics are the main problems
* IQ>80
* If medication, then has been stable for at least one months in medicated patients
* No change in medication treatment is planned
* Ability to participate in weekly outpatient treatment
* Acceptance of randomization

Exclusion Criteria:

* Diagnosis of Autism Spectrum Disorder or Psychosis
* Parallel continuous psychotherapy of tics or comorbid

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-11; Primary Completion 2017-06 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Change in Symptom Checklist for Tic-Symptoms (FBB-TIC), parent rating | Baseline (T0), after 8 weeks (T1), 16weeks (T2), 24weeks (T3)
  The FBB-TIC is used to assess Tic-Symptoms according to DSM-IV and ICD-10 rated by parents
Change in self-esteem (Harter-Scale-SBB)(self rating) | T0, after 8 weeks (T1), 24weeks (T3)
  The Harter-Scale is used to assess self-esteem

SECONDARY OUTCOMES:
Change in Symptom Checklist for Tic-Symptoms (FBB-/SBB-TIC), Teacher-/self-rating | Baseline (T0), after 8 weeks (T1), 16 weeks (T2), 24weeks (T3)
  The SBB-TIC is used to assess Tic-Symptoms according to DSM-IV and ICD-10 rated by parents
Change in Symptom Checklist for Tic-Symptoms, clinical rating | Baseline (T0), after 8 weeks (T1), 16weeks (T2), 24weeks (T3)
  The Checklist is used to assess Tic-Symptoms according to DSM-IV and ICD-10 rated by clinicians
Change of comorbid ADHD Symptoms (FBB/SBB-ADHD), parent, teacher and self-rating | T0, after 8 weeks (T1), 24 weeks (T3)
  The Symptom Checklist for Attention Deficit/Hyperactivity Disorder (FBB-/SBB-ADHS) assess all symptom criteria according to DSM IV and ICD-10.
Change of comorbid OCD Symptoms (ZWIK-E), parent-rating | T0, after 8 weeks (T1), 24weeks (T3)
  The ZWIK assess OCD criteria.
Change of comorbid Symptoms (CBCL/TRF/YSR), parent-/teacher-/self-rating | T0, after 8 weeks (T1), 24weeks (T3)
  The CBCL, TRF and YSR assess a variation of different criteria.
Change in Tic-Symptoms (YGTSS-TIC), overall score | Baseline (T0), after 8 weeks (T1),16weeks (T2), 24weeks (T3)
  The YGTSS is used to assess Tic-Symptoms in a semi structured interview with parents and patients
Change in Tic-Symptoms (observation) | Between T1 and T3 up to 16 weeks, during each session/week
  Tic symptoms are observed through video tapes and are rated through clinicians

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Döpfner, Prof. Dr., Study Director — Department of Childhood and Adolescent Psychiatry and Psychotherapy
Locations (1):
- University Hospital of Cologne, Department of Childhood and Adolescent Psychiatry and Psychotherapy, Cologne, Germany

REFERENCES:
- [Background] Perri, D., Mandler, J. & Döpfner, M. (2015). STARK - Supportive Therapie zur Aktivierung von Ressourcen. Göttingen: Hogrefe.